CLINICAL TRIAL: NCT07394140
Title: Evaluate Functionality and Use of the NMT EasyFit Sensor and NMT EasyFit Cable
Brief Title: NMT EasyFit Sensor and Cable
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SA-000175
Record Dates: First submitted 2026-02-02; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Neuromuscular Blockade Monitoring; Neuromuscular Monitoring After Administration of Neuromuscular Blocking Agents in Different Types of Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- All Subjects (Experimental): Placement of NMT Sensor
  Interventions: Device: NMT Technology

INTERVENTIONS:
Device: NMT Technology — Collection and assessment of non-invasive electrical stimuli from the NMT measurement placed on the patient's hand and forearm to measure the level of neuromuscular blocking agents during standard of care surgical procedures.

SUMMARY:
The purpose of this clinical study is to collect and assess feedback from clinical users regarding the functionality and device use and collection of raw parameter date from the NMT Sensor and NMT Cable.

DETAILED DESCRIPTION:
The NMT Sensor provides quantitative, automated measurements of neuromuscular block by delivering non-invasive electrical stimuli to the ulnar nerve and recording electromyography (EMG) responses from the adductor pollicis muscle. Surface hydrogel electrodes with adhesive foam ensure secure placement for continuous monitoring. The single-use sensor connects to a reusable NMT Cable and is designed for use with GE HealthCare NMT measurement devices (NMT Module and bedside monitors).

ELIGIBILITY:
Inclusion Criteria:

1. Study subject (male or female) is age 18 years or older (≥18 years).
2. Study subject must have the ability to understand and provide written informed consent.
3. Study subject is undergoing a clinically indicated procedure requiring the use of paralytic medication.
4. Study subject will have the primary NMT monitoring conducted using an NMT ElectroSensor on the hand/forearm.

Exclusion Criteria:

1. Are known to be pregnant.
2. Are breastfeeding.
3. Suffering from an infection(s) that requires isolation.
4. Deformity, scar tissue, tattoos, or other characteristics at the sensor application area that could interfere (e.g., nerve damage) with the completion of the study procedure or identify a study subject.
5. Subjects requiring rapid sequence induction
6. Subjects expected to be at risk from participation for any reason, such as those with known allergy or sensitivity to adhesive materials that may be used in the study.
7. Direct employees or contractors of GE HealthCare, or any company that makes NMT monitoring devices (sensors, cables, modules).
8. NMT ElectroSensor placed on the foot/ankle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Collection of End User Feedback Surveys | Up to 24 hours
  Collection of end user feedback surveys on the functionality and clinical use of the NMT Sensor and Cable during standard of care surgical procedure (minimum of 1 hour and maximum of 24 hours).

SECONDARY OUTCOMES:
Collection of raw parameter data from NMT Sensor and Cable | Up to 24 hours
  Collection of raw parameter data from NMT Sensor and Cable to evaluate the reliability of the measurements to NMBA concordance rate.
Incidence of Safety Events | 4 months.
  Analysis of adverse events will be listed per subject, summarized with counts and percentages of events, and summarized with counts and percentages of subjects with events.

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States